CLINICAL TRIAL: NCT01008527
Title: A Phase I Study of Poly IC:LC and NY-ESO-1/gp100 Peptides Either Emulsified With Montanide ISA 51 or in Aqueous Solution With Escalating Doses of CP 870,893 in the Treatment of Subjects With Resected Stage III or Stage IV Melanoma
Brief Title: Phase I Oncovir Poly IC:LC and NY-ESO-1/gp100
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oncovir, Inc. (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15383; 106566 (Other: USF IRB); NCI-P-8215 (Other: NCI)
Record Dates: First submitted 2009-11-02; First posted 2009-11-05 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Melanoma
Keywords: skin; cutaneous; immunotherapy; immunology; dose escalation
MeSH Terms: conditions — Melanoma | interventions — selicrelumab; Peptides; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infusion and Peptide Administration (Experimental): Patients get the study drug Oncovir poly IC:LC with or without CP 870-893. Up to 6 groups of 3 to 10 patients each will be treated in this study. The first group (between 3 and 6 patients) gets peptide vaccine with poly IC:LC. Second, third and fourth groups of 3 to 6 patients receive peptide vaccine with poly IC:LC and the antibody CP 870,893 at increasing doses from 0.01, 0.025 and 0.05 mg/kg. CP 870-893 will be given to 10 patients at a dose of 0.1 mg/kg to patients in the fifth group, and 0.2 mg/kg to the sixth group. The CP 870,893 will be given as an intravenous infusion over 30 minutes and will be given once every 2 weeks for the first 6 infusions. CP-870-893 will then be given every 4 to 6 weeks for 3 injections. The final 3 injections of CP 870,893 will be given every 8 to 12 weeks. These infusions will take place on weeks 1, 3, 5, 7, 9, 11, 17, 21, 25, 33, 41, and 53 for a total of 12 infusions.
  Interventions: Drug: CP 870,893; Biological: Peptides; Biological: Oncovir poly IC:LC

INTERVENTIONS:
Drug: CP 870,893 — Study drug will be administered open-label as an intravenous solution, followed by observation. Study drug will be supplied as a liquid intravenous solution in vials containing 10 mg/mL of CP870,893. CP 870,893 will be administered at a dosage of 0.01, 0.025 or 0.05 mg/kg at 0.24 mg/mL infused via a syringe pump over 15 minutes, or at 0.1 or 0.2 mg/kg/dose as an i.v. infusion in saline at a concentration of 0.24 mg/mL in an IV bag of up to 100 mL over 30 minutes (controlled by a volumetric pump) for not more than 30 minutes, with a 10 cc flush at the end that should be administered at the same rate as the CP 879,893 infusion.
  Other Names: NSC 750268
Biological: Peptides — NY-ESO-l 157-165 (165V) and gpl002 80-288 (288V) peptides each at a dose of 0.5 mg will be emulsified with Montanide ISA 51 VG and administered to all patients in the study at Weeks 1,3, 5, 7, 9, 11, 17, 21, 25 33, 41, and 53. Peptides will be administered as a total of 6 deep subcutaneous (s.c.) injections into alternating lower extremities one hour after CP 870,893 infusions.
  Other Names: NSC 717388; NSC 683473; NSC 737063
Biological: Oncovir poly IC:LC — The dosage of poly IC:LC chosen for the current trials has been used safely in over one hundred patients with central nervous system (CNS) malignancies enrolled in nitrates and bone turnover (NABT) trials. The injection of 1000 mcg will be made deeply subcutaneously into the same limb as the peptides/Montanide ISA 51 VG, at least 5 cm. proximal to the peptides vaccination site. Poly IC:LC will be administered to all patients in the study at Weeks 1, 3, 5, 7, 9, 11, 17, 21, 25 33, 41, and 53 one hour after CP 870,893 infusion.
  Other Names: Hiltonol; NSC 301463

SUMMARY:
The purpose of this study is to determine what side effects CP 870,893 may cause when given with an immune stimulant called Oncovir poly IC:LC along with a melanoma vaccine. The CP 870,893, the Oncovir poly IC:LC and the melanoma vaccine are investigational drugs that have not been combined in patients before, and that have not been approved for sale by the Food and Drug Administration. The Oncovir poly IC:LC is intended to stimulate the body's immune system.

DETAILED DESCRIPTION:
Antibodies such as CP 870,893 are chemicals made by immune cells naturally found in the human body. CP 870,893 was produced in cells grown from a hamster but is fully human in composition. The vaccine contains peptides (pieces) from two different proteins called NY-ESO-1 and gp100. Each one is made by 50-100% of melanomas. These proteins can be recognized by the immune system. They will be injected under the skin of the participant's thigh in combination with, or without an oil-based substance, called "Montanide ISA 51 VG". The Montanide ISA 51 VG is an adjuvant or "assistant" which stimulates the body's immune system. The peptides in the vaccine, the Montanide ISA 51 VG, the Oncovir poly IC:LC and the CP 870,893 antibody are not approved by the Food and Drug Administration (FDA) but the FDA is permitting their use in this study. It is believed that the CP 870,893 and the Oncovir poly IC:LC will boost the body's immune response against the melanoma vaccine, although this vaccine has not been proven to help the patient's melanoma.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria on pre-study examination (within 28 days prior to study drug administration) to be eligible to participate in the study:

* Have read, understood, and provided written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization after the nature of the study has been fully explained
* Histologic diagnosis of Stage III (with ≥ 3 positive lymph nodes) or Stage IV melanoma that has been resected completely (may include mucosal or ocular melanoma) no more than 6 months prior to screening
* Human leukocyte antigen (HLA)-A*0201 status as determined by deoxyribonucleic acid (DNA) allele-specific polymerase chain reaction (PCR) assay
* Positive staining of tumor tissue with at least one of the following: antibody HMB-45 for gplOO, NY-ESO-l, or MART-I
* At least 4 weeks since treatment (surgery, chemotherapy, immunotherapy, radiotherapy) and at least 6 weeks for treatment with nitrosoureas for melanoma, and at least 8 weeks since adjuvant treatment with an anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody for melanoma and recovered from any serious toxicity experienced during treatment
* Women must be either: post-menopausal for at least 1 year; surgically incapable of bearing children; or utilizing a reliable form of contraception during the study and for at least 4 months after the final CP 870,893 infusion or vaccination. Women of childbearing potential must have a negative serum hCG- ß pregnancy test conducted during the screening period and have a negative urine pregnancy test conducted on the day of each infusion (prior to the infusion).
* Men who may father a child must agree to the use of male contraception for the duration of their participation in the trial and for at least 4 months after the final CP 870,893 infusion or vaccination.
* Patients with Stage III resected melanoma rendered free of disease can have failed treatment with, been ineligible for, or refused treatment with a-interferon.
* Analgesic therapy must be stable for a period of 14 days prior to infusion of study drug.
* Life expectancy ≥ 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients with resected brain metastases that are off steroids, have no evidence of disease by brain magnetic resonance imaging (MRI) scanning, or computer tomography (CT) of the brain if an MRI cannot be performed, are eligible.
* Screening laboratory values must meet the following criteria: white blood cell (WBC): ≥2500 cells/mm³; absolute neutrophil count (ANC): ≥1500 cells/mm³, Platelets: ≥100,000/mm³; Hematocrit: ≥30%; Hemoglobin: ≥10 g/dL; Creatinine: ≤2.0 mg/dL; aspartate aminotransferase (AST): ≤3 x ULN; Bilirubin: ≤1.0 x upper limit of normal (ULN) (except patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dL); human immunodeficiency virus (HIV): negative; HBsAg: negative; hepatitis C virus (HCV) antibody [anti-HCV Ab]: nonreactive. If reactive, patient must have a negative HCV RNA qualitative PCR.

Exclusion Criteria:

* Any prior malignancy except for the following: adequately treated basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix, or any other cancer from which the patient has been disease-free for at least 5 years.
* History of any autoimmune disease, specifically including the following diseases: inflammatory bowel disease or any other autoimmune bowel diseases; systemic lupus erythematosis; rheumatoid arthritis; or any autoimmune ocular diseases. Patients with an autoimmune disease history affecting the pancreas, pituitary, liver, gastrointestinal (GI) tract or adrenals, and prior history of Guillan-Barre and other neurologic conditions felt to be autoimmune in nature are also excluded.
* Active infection, requiring therapy, chronic active hepatitis B virus (HBV) or HCV, or confirmed reactivity with HIV tests.
* Pregnancy or nursing: due to the possibility that CP 870,893 could have a detrimental effect on the developing immune system of the fetus or infant, exposure in utero or via breast milk will not be allowed.
* Systemic hypersensitivity to Montanide ISA 51 (IFA), Montanide ISA 51 VG or any vaccine component
* Any underlying medical condition which, in the opinion of the Principal Investigator (PI), will make the administration of study drug hazardous or obscure the interpretation of adverse events.
* Any concurrent medical condition requiring the use of systemic, inhaled or topical corticosteroids or the use of immunosuppressive agents (e.g. cyclosporine and its analog, or chemotherapy agents). All corticosteroid use must have been discontinued at least 4 weeks prior to study entry.
* Prior treatment with CP 870,893 or any anti-CD40 antibody
* Evidence or history of significant cardiac, pulmonary, hepatic, renal, psychiatric or gastrointestinal disease that would make the administration of CP 870,893 unsafe
* Concurrent treatment with chemotherapy or other immunotherapy regimens (must be completed at least 4 weeks before Screening; 6 weeks for nitrosoureas); prior treatment with chemotherapy, radiotherapy or other than anti CD40 antibodies will not be an exclusion.
* History of prior allogeneic human stem cell or bone marrow transplant
* History of prior thromboembolic venous events, or inherited / acquired coagulopathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2013-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 3 Years
  The overall goal is to define a safe and potentially effective dose and schedule of CP 870,893 with Oncovir poly IC:LC with a peptide vaccine with either Montanide ISA 51 VG or in aqueous solution for the adjuvant setting in high risk melanoma.

SECONDARY OUTCOMES:
Number of Participants With Immunologic Response | 3 Years or until relapse
  To assess immune responses to the study regimens.
Number of Participants With Progression Free Survival (PFS) | 3 Years or until relapse
  Relapse free survival will be summarized in a standard exploratory fashion via descriptive summary statistics by dose.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weber, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States